CLINICAL TRIAL: NCT01884636
Title: A Phase 1, Open- Label Study to Evaluate the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of Methotrexate
Brief Title: A Study to Evaluate the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of Methotrexate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0052
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Methotrexate; Pharmacokinetics of 7-hydroxymethotrexate; Healthy Subjects
Keywords: Isavuconazole; Pharmacokinetics; Healthy Subjects; BAL8557; BAL4815; methotrexate
MeSH Terms: interventions — isavuconazole; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- isavuconazole and methotrexate (Experimental): Methotrexate single dose on days 1 and 8. Isavuconazole three times a day (TID) on days 4 and 5 followed by isavuconazole once daily (QD) on days 6 - 9
  Interventions: Drug: isavuconazole; Drug: methotrexate

INTERVENTIONS:
Drug: isavuconazole — oral
  Other Names: BAL8557
Drug: methotrexate — oral

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics of a single dose of methotrexate. Safety and tolerability of isavuconazole will be assessed alone and in combination with methotrexate.

DETAILED DESCRIPTION:
Subjects will check-in to the clinic on Day -1 and remain confined through completion of the study procedures on Day 10.

A follow-up telephone call will be made on Day 16 to check on health status.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and a body mass index of 18 to 32 kg/m2, inclusive.
* QTcF must be 360 to 430 msec.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and serum creatinine must not be above the normal range.
* Male subject must be using highly effective contraception from Screening through 90 days after final study drug administration.
* Male subject must not donate sperm starting at Screening through 90 days after final study drug administration.

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of either Short or Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes).
* The subject has a history of tuberculosis, or has a known or suspected immunodeficiency syndrome.
* The subject has a positive result for hepatitis B surface antigen, hepatitis C antibodies or QuantiFERON®-TB Gold test(s) at Screening or is known to be positive for human immunodeficiency virus.
* The subject has a known or suspected allergy to any of the components of the trial products or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods, or a history of severe anaphylactic reactions.
* The subject is a smoker (any use of tobacco or nicotine containing products) in the last 6 months.
* The subject has had treatment with any prescribed or non-prescribed drugs in the 2 weeks prior to Day 1, with the exception of occasional use of acetaminophen up to 2 g/day.
* The subject has participated in any interventional clinical study or has received any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to Screening.
* The subject has participated in a prior study with isavuconazole.
* The subject has history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening or the subject tests positive at screening or Day -1 for alcohol or drugs of abuse.
* The subject is an employee of the Astellas Group or vendors involved in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of methotrexate in plasma: Area Under the Concentration-Time Curve (AUC) from the time of dosing to the last quantifiable concentration (AUClast) | Days 1 and 8 (15 plasma samples obtained from time zero to 36 hours post dose)
PK of methotrexate in plasma: AUC from the time of dosing to infinity (AUCinf) | Days 1 and 8 (15 plasma samples obtained from time zero to 36 hours post dose)
PK of methotrexate in plasma: Maximum Concentration (Cmax) | Days 1 and 8 (15 plasma samples obtained from time zero to 36 hours post dose)

SECONDARY OUTCOMES:
PK variable for isavuconazole in plasma: Trough Concentration (Ctrough) | Days 6, 9 and 10 (1 sample prior to isavuconazole dosing)
Composite of PK variables for isavuconazole in plasma: AUCtau, Cmax and tmax | Days 7 and 8 (13 samples collected per day)
  AUC during the time interval between consecutive dosing (AUCtau); the time after dosing when Cmax occurs (tmax)
Composite of PK variables for methotrexate in plasma: t1/2, tmax, CL/F and Vz/F | Days 1 and 8 (15 plasma samples obtained from time zero to 36 hours post dose)
  Apparent Terminal Elimination Half-life (t1/2); Apparent Body Clearance After Oral Dosing (CL/F); Apparent Volume of Distribution (Vz/F)
Composite of PK variables for 7- hydroxymethotrexate in plasma: AUClast, AUCinf, t1/2, Cmax and tmax | Days 1 and 8 (15 plasma samples obtained from time zero to 36 hours post dose)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States